CLINICAL TRIAL: NCT02321449
Title: Open-label, Post-marketing Observational Study to Evaluate the Effectiveness of Circadin in Improving Quality of Sleep in Patients Aged 55 or Over
Brief Title: The Effectiveness of Circadin in Improving Quality of Sleep in Patients Aged 55 or Over
Acronym: QUALISLEEP
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-38-59010-001
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate the effectiveness of treatment with Circadin based on sleep improvement as assessed by the modified Questionnaire Scoring Subjective Characteristics of Sleep before and after the treatment

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged ≥ 55 years suffering from non-organic insomnia according to International Classification of Diseases (ICD-10)
* Patients with sleep disorders manifested as poor sleep quality associated with impaired daytime functioning with or without one or more of the following criteria: difficulty falling asleep, frequent night awakenings, early morning awakenings
* Patients able to follow the study protocol
* Patients who have signed the Informed Consent prior to initiation of any observation-related procedures
* Patients with a global score of ≤17 inclusively on the modified Questionnaire Scoring Subjective Characteristics of Sleep
* Patients who have just been identified to receive treatment with Circadin
* Patients without previous treatment with Circadin

Exclusion Criteria:

* Hypersensitivity to any components of Circadin
* Congenital galactose intolerance, glucose-galactose malabsorption, Lapp lactase deficiency
* Pregnancy and lactation
* Alcohol or drug addiction
* Severe somatic and neurological conditions, exacerbations thereof, including autoimmune diseases or renal/hepatic insufficiency
* Intake of psychoactive medicines within the last 30 days before observational study entry
* Presence of clinically significant anxiety and depression as assessed by the Hospital Anxiety and Depression Scale
* Presence of pain that might be the cause for insomnia. Subjects suffering from breathing related sleep disorders

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male and female patients aged ≥ 55 years suffering from primary (non-organic) insomnia characterized by poor quality of sleep
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in quality of sleep questionnaire | Baseline, 3 weeks
  Sleep improvement as assessed by the modified Questionnaire Scoring Subjective Characteristics of Sleep before and after treatment.

SECONDARY OUTCOMES:
Change from baseline in attention Questionnaire | Baseline, 3 weeks
Change from baseline in memory Questionnaire | Baseline, 3 weeks
Percentage of patients responding "unsatisfied", "effective therapy", "very effective therapy", respectively, in the patient satisfaction assessment | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (3):
- Russia (3):
  - State research center of preventive medicine, Moscow
  - Research and Education Center of Moscow State University named after M.V. Lomonosov, Moscow
  - First Moscow State Medical University, Moscow